CLINICAL TRIAL: NCT01967810
Title: A Phase II, Open-Label, Multi-Center Study of ANG1005 in Patients With Recurrent High-Grade Glioma
Brief Title: ANG1005 in Patients With Recurrent High-Grade Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Angiochem Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANG1005-CLN-03
Record Dates: First submitted 2013-10-09; First posted 2013-10-23 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Glioma; Glioblastoma; Brain Tumor, Recurrent
Keywords: glioma; glioblastoma; brain cancer; brain tumor; recurrent
MeSH Terms: conditions — Glioma; Glioblastoma; Brain Neoplasms; Recurrence | interventions — paclitaxel-Angiopep-2 conjugate; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Experimental): ANG1005 administered to bevacizumab-naive recurrent GBM participants
  Interventions: Drug: ANG1005
- Arm 2 (Experimental): ANG1005, with or without bevacizumab, administered to bevacizumab-refractory recurrent GBM participants
  Interventions: Drug: ANG1005; Drug: Bevacizumab
- Arm 3 (Experimental): ANG1005 administered to recurrent WHO Grade III anaplastic glioma participants
  Interventions: Drug: ANG1005

INTERVENTIONS:
Drug: ANG1005 — ANG1005 at a starting dose of 650 mg/m^2 or 600 mg/m^2 by intravenous infusion once every 3 weeks
  Other Names: GRN1005
Drug: Bevacizumab — For participants enrolled in the bevacizumab-refractory recurrent GBM arm (Arm 2), treatments with bevacizumab may be continued and administered every 2 or 3 weeks at the Investigator's discretion.
  Other Names: Avastin
  Arms: Arm 2

SUMMARY:
This is a Phase 2 study to see if an investigational drug, ANG1005, can shrink tumor cells in patients with high-grade glioma. Another purpose of this study is to assess the efficacy, safety, tolerability, and pharmacokinetics (PK) of ANG1005 in patients.

DETAILED DESCRIPTION:
See above.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years old
2. GBM and GBM variants, WHO Grade III anaplastic glioma diagnosis confirmed
3. Radiologically confirmed recurrent and bi-dimensionally measurable disease per Response Assessment in Neuro-Oncology (RANO) criteria
4. Neurologically stable
5. For bevacizumab-refractory patients, radiologic demonstration of tumor progression during bevacizumab therapy
6. Karnofsky performance status (KPS) ≥ 80
7. Expected survival of at least 3 months

Exclusion Criteria:

1. More than three relapses
2. Previous ANG1005/GRN1005 treatment
3. Radiotherapy within 3 months.
4. Therapy with bevacizumab within 4 weeks prior to Day 1 of treatment for recurrent WHO grade III anaplastic glioma patients (Arm 3)
5. Evidence of significant intracranial hemorrhage
6. Previous taxane treatment
7. Prior therapy with bevacizumab for bevacizumab-naïve patients (Arm 1)
8. NCI Common Toxicity Criteria for Adverse Effects (CTCAE) v4.0 Grade ≥ 2 neuropathy
9. Inadequate bone marrow reserve
10. Any evidence of severe or uncontrolled diseases
11. Participants with the presence of an infection including abscess or fistulae, or known infection with hepatitis C or B or HIV
12. Known severe hypersensitivity or allergy to paclitaxel or any of its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2013-10; Primary Completion 2016-02 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) (Arms 1 and 3) | Upon enrollment through end of study period (1 year after last patient is enrolled)
  To determine the radiologic ORR in bevacizumab-naïve recurrent Glioblastoma multiforme (GBM) patients (Arm 1)and in recurrent anaplastic glioma World Health Organization (WHO) Grade III patients (Arm 3)
PFS3 (Arm 2) | Upon enrollment through end of study period (1 year after last patient is enrolled)
  To determine the progression-free survival at 3 months (PFS3) in bevacizumab-refractory recurrent GBM patients (Arm 2)

SECONDARY OUTCOMES:
ORR in Arm 2 | Upon enrollment through end of study period (1 year after last patient is enrolled)
  To determine the ORR in Arm 2
PFS at 3, 6 and 12 months | Upon enrollment through end of study period (1 year after last patient is enrolled)
  * To determine the number of patients without progression at 3, 6 and 12 months in Arms 1 and 3
  * To determine the number of patients without progression at 6 and 12 months in Arm 2
Median PFS | Upon enrollment through end of study period (1 year after last patient is enrolled)
  To determine the median progression-free survival in each arm
Duration of response | Upon enrollment through end of study period (1 year after last patient is enrolled)
  To determine the median duration of response in each arm
Overall survival | Upon enrollment through end of study period (1 year after last patient is enrolled)
  To determine the median overall survival in each arm
Safety and tolerability | Upon enrollment through end of study period (1 year after last patient is enrolled)
  To determine the number of participants with adverse events
Plasma Pharmacokinetics of ANG1005 (Half-life [T1/2], Maximum Concentration [Cmax], Area Under the Curve [AUC]) | At 0 h (pre-dose), at the end of infusion, at 2 and 4 hours post-dose on Day 1 of treatment cycles 1 and 3 (Week 1 and Week 9)
  To determine the drug concentration and distribution in the blood (plasma)

CONTACTS AND LOCATIONS:
Overall Officials: Betty Lawrence, Study Director — Angiochem Inc
Locations (12):
- United States (12):
  - Moores UC San Diego Cancer Center, La Jolla, California
  - Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Cleveland Clinic, Cleveland, Ohio
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Univeristy of Texas Health Science Center in San Antonio, San Antonio, Texas
  - Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Dmello C, Brenner A, Piccioni D, Wen PY, Drappatz J, Mrugala M, Lewis LD, Schiff D, Fadul CE, Chamberlain M, Kesari S, Ahluwalia M, Ghosh D, Sonabend AM, Kumthekar P. Phase II trial of blood-brain barrier permeable peptide-paclitaxel conjugate ANG1005 in patients with recurrent high-grade glioma. Neurooncol Adv. 2024 Dec 14;6(1):vdae186. doi: 10.1093/noajnl/vdae186. eCollection 2024 Jan-Dec. PMID 39713041
- See also: A Phase I sudy of ANG1005 (GRN1005) in recurrent malignant glioma — http://www.ncbi.nlm.nih.gov/pubmed/23349317